CLINICAL TRIAL: NCT02082418
Title: Effects of Alpha-lactalbumin on Metabolic and Cognitive Functions in Healthy Older Adults
Brief Title: Effects of Alpha-lactalbumin Intake on Metabolic and Cognitive Functions in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-0065
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild cognitive impairment; Protein digestion; Tryptophan digestion; Cognitive function; Mood; Muscle function; Alpha-lactalbumin
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Lactalbumin; Whey; Caseins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy (Experimental): healthy control subjects
  Interventions: Dietary Supplement: Alpha-lactalbumin; Dietary Supplement: Whey; Dietary Supplement: Casein
- MCI (Experimental): mild cognitive impariments
  Interventions: Dietary Supplement: Alpha-lactalbumin; Dietary Supplement: Whey; Dietary Supplement: Casein
- Dementia (Experimental): established diagnosis of dementia
  Interventions: Dietary Supplement: Alpha-lactalbumin; Dietary Supplement: Whey; Dietary Supplement: Casein

INTERVENTIONS:
Dietary Supplement: Alpha-lactalbumin — Subjects will ingest the liquid meal containing alpha-lactalbumin and carbohydrates (0.6 g/kg FFM protein + 0.3 g/kg FFM carbohydrates).
Dietary Supplement: Whey — commercially available whey protein
Dietary Supplement: Casein — commercially available casein protein

SUMMARY:
Aging modifies the metabolic pathway of the neurotransmitter serotonin by reducing the synthesis rate and increasing the breakdown rate of serotonin, possibly related to the observed enhanced sensitivity of the serotonergic pathway. Since serotonin plays a prominent role in neuropsychological functions such as anxiety, mood and memory, the enhanced sensitivity of the serotonergic pathway in aging can probably explain the fact that elderly are more vulnerable to develop cognitive deficits and depressive symptoms.

Serotonin synthesis in brain is regulated by its precursor tryptophan (TRP). Because tryptophan is an essential amino acid, modifying the availability of tryptophan through dietary intake, can directly influence central serotonin metabolism and consequently affective and cognitive processes.

The aim of this study is to test the hypothesis that an acute intake of whey protein with high levels of TRP such as alpha-lactalbumin can stabilize the metabolism of serotonin and subsequently enhance metabolic and cognitive functions in healthy older adults. The acute effects of this dietary protein will be investigated in subjects with mild cognitive impairment (MCI), or dementia, compared to control subjects in order to examine whether healthy older subject with MCI benefit more from the intake of alpha-lactalbumin and/or whey. The investigators will investigate if this meal can optimize serotonin metabolism by elevating plasma TRP levels and plasma TRP appearance and enhance splanchnic TRP extraction. In addition, the effects on mood and cognitive functions will be examined.

DETAILED DESCRIPTION:
The study involves for all subjects 3 test days (approximately 8 hours each). On this test day the investigators will examine the acute effects of a protein meal. Subjects will receive a mixture of alpha-lactalbumin and/or whey and/or casein, carbohydrates and amino acid stable isotopes to investigate protein and amino acid kinetics (assigned to alpha-lactalbumin or whey or casein group on test day 1, then switch on test day 2 and 3). The subjects will receive these stable isotopes by infusion in their blood and by oral intake (e.g. simultaneously with protein meal). For study purposes, blood will be drawn approx. 25 times during 8 hours on the test day, altogether about 100-120 ml of blood will be drawn on the test day.

ELIGIBILITY:
Inclusion criteria subjects with dementia:

* Dementia diagnosis
* Ability to walk, sit down and stand up independently
* Age 55 years or older
* Ability to lie in supine or elevated position for 8 hours
* Willingness and ability to comply with the protocol, including:

Adhering to fasting state from 10 pm ± 2h onwards the day prior to each study visit

Inclusion criteria healthy subjects:

* Healthy male or female according to the investigator's or appointed staff's judgment
* Ability to walk, sit down and stand up independently
* Age 55 years or older
* Ability to lie in supine or elevated position for 8 hours
* Willingness and ability to comply with the protocol, including:

Adhering to fasting state from 10 pm ± 2h onwards the day prior to each study visit

Exclusion Criteria:

* Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (for healthy control group only)
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* Indication of severe cognitive impairment (MOCA score < 17)
* Established diagnosis of Insulin Dependent Diabetes Mellitus
* History of untreated metabolic disease(s) including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Presence of fever within the last 3 days
* Preplanned surgery of procedures that would interfere with the conduct of the study
* Any other condition according to the PI or study physician that would interfere with proper conduct of the study / safety of the patient
* Current alcohol or drug abuse
* Known allergy to milk or milk products
* Use of long-term oral corticosteroids or short course of oral corticosteroids 4 weeks preceding first test day
* Use of protein or amino acid containing nutritional supplements within 5 days of test day
* (Possible) pregnancy
* BMI of < 18.5 or ≥ 40 kg/m2
* Dietary or lifestyle characteristics: When during the period from enrollment to completion of the study (end of test day) any condition is developed, whether causing the subject to not meet inclusion criteria or to meet exclusion criteria, the subject will be excluded from the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Net whole-body protein synthesis | 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210 min post-meal
  Change in whole-body protein synthesis rate after intake of meal

SECONDARY OUTCOMES:
Citrulline rate of appearance | Postabsorptive state during 2 hours
  Plasma enrichment of citrulline
Skeletal and respiratory muscle strength | 1 day
  Difference in leg strength and fatigue, handgrip strength and fatigue, and inspiratory and expiratory pressure between older adults with and without MCI.
Cognitive function and mood | Postabsorptive state during 3 hours and change after feeding
  Outcome of neuro-psychological tests in healthy older adults with and without MCI in relation to the tryptophan metabolism
Protein digestion after feeding | 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210 min post-meal
  Ratio enrichment free phenylalanine versus phenylalanine from protein spirulina
Arginine turnover rate | Postabsorptive state during 3 hours
  Arginine enrichment in plasma
Whole body collagen breakdown rate | Postabsorptive state during 3 hours
  Hydroxyproline enrichment in plasma
Tryptophan turnover rate | Postabsorptive state during 3 hours and change after feeding
  Tryptophan enrichment in plasma in postabsorptive state and after intake of meal
Insulin response to feeding | During 3 hours after feeding
  Acute change from postabsorptive state after intake of meal
Fat-free mass | Postabsorptive state during 15 min
  Characteristics of study subjects
Myofibrillar protein breakdown rate | 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210 min post-meal
  3methylhistidine enrichment in plasma
Glycine rate of appearance | Postabsorptive state during 3 hours
  Glycine enrichment in plasma
Taurine turnover rate | Postabsorptive state during 3 hours
  Enrichment of taurine in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Marielle P Engelen, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

REFERENCES:
- [Derived] Yu AK, Deutz NEP, Perez CN, DeWandel S, Ruebush LE, Engelen MPKJ. The acute effects of alpha-lactalbumin intake on tryptophan metabolites and mood in older adults with Mild Cognitive Impairment. Nutr Neurosci. 2025 Sep 14:1-15. doi: 10.1080/1028415X.2025.2554359. Online ahead of print. PMID 40946231
- [Derived] Deutz LN, Wierzchowska-McNew RA, Deutz NE, Engelen MP. Reduced plasma glycine concentration in healthy and chronically diseased older adults: a marker of visceral adiposity? Am J Clin Nutr. 2024 Jun;119(6):1455-1464. doi: 10.1016/j.ajcnut.2024.04.008. Epub 2024 Apr 12. PMID 38616018